CLINICAL TRIAL: NCT00515385
Title: A Phase 1, Randomized, Double-Blind, Dose-Escalation Cohort Study to Evaluate the Safety, Tolerability and Pharmacokinetics of a Single Intravenous Infusion of MGAWN1, a Neutralizing, Humanized, Monoclonal Antibody (IgG1k) to West Nile Virus, in Healthy Adults
Brief Title: A Trial to Evaluate the Safety of a Single Intravenous Infusion of MGAWN1 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-MGAWN1-01; DMID 06-0090
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: West Nile Virus
Keywords: Randomized; Double-Blind; Dose-Escalation; Cohort Study

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (10):
- 1a (Experimental): Cohort 1 completed
  Interventions: Drug: MGAWN1
- 1b (Placebo Comparator): Cohort 1 placebo completed
  Interventions: Drug: MGAWN1; Other: Placebo
- 2a (Experimental): Cohort 2 completed completed
  Interventions: Drug: MGAWN1
- 2b (Placebo Comparator): Cohort 2 placebo completed
  Interventions: Drug: MGAWN1; Other: Placebo
- 3a (Experimental): Cohort 3 active
  Interventions: Drug: MGAWN1
- 3b (Placebo Comparator): Cohort 3 placebo
  Interventions: Drug: MGAWN1; Other: Placebo
- 4a (Experimental): Cohort 4 active
  Interventions: Drug: MGAWN1
- 4b (Placebo Comparator): Cohort 4 placebo
  Interventions: Drug: MGAWN1; Other: Placebo
- 5a (Experimental): Cohort 5 active
  Interventions: Drug: MGAWN1
- 5b (Placebo Comparator): Cohort 5 placebo
  Interventions: Drug: MGAWN1; Other: Placebo

INTERVENTIONS:
Drug: MGAWN1 — Eight subjects per cohort, each receives a single IV infusion of MGAWN1 of saline control on study day 0 (6 MGAWN1, 2 saline control.
  Cohort 1 - 0.3 mg/kg Cohort 2 - 1 mg/kg Cohort 3 - 3 mg/kg Cohort 4 - 10 mg/kg Cohort 5 - 30 mg/kg
Drug: MGAWN1 — Single IV dose
  Arms: 1a; 2a; 3a; 4a; 5a
Other: Placebo — Single IV dose
  Arms: 1b; 2b; 3b; 4b; 5b

SUMMARY:
The primary purpose of this phase 1, double-blind, cohort study is to evaluate the safety, tolerability, and pharmacokinetics of escalating doses of MGAWN1 administered as a single intravenous (IV) infusion to healthy adults. Subjects will be enrolled sequentially into one of 5 dose-level cohorts, with 8 subjects in each cohort. Six subjects in each cohort will receive MGAWN1 (a Neutralizing, Humanized, Monoclonal Antibody (IgG1k) to West Nile Virus) and 2 will receive a saline control.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the subject including consent for the use of research-related health information, before performance of any study-related procedure including screening procedures
2. Healthy adult male or female subjects aged 18-65 years, with a body mass index (BMI) of 18-32 kg/m2
3. Subjects must be physically healthy as determined by the investigator based on medical history, physical examination, ECG, and clinical laboratory tests within laboratory normal ranges. To be considered normal, the following results must pertain:

   * The serum potassium must be within normal limits.
   * Hemoglobin must be ≥12 mg/dl; ANC must be 1,500-upper limit of normal (ULN); platelets must be 130,000-500,000 μL; and sodium must be 130-150 moles/L.
   * Each of these tests must not exceed the upper limit of normal: WBC, creatinine, and (provided asymptomatic) fasting blood glucose.
   * Bilirubin must be ≤ 2x ULN, ALT ≤ 1.25x ULN, and AST ≤1.25x ULN
   * Urinalysis: glucose negative and protein ≤ 20 mg/dl.
4. Have adequate venous access
5. Have negative assays for human immunodeficiency virus (HIV), hepatitis B virus (HBsAg) and hepatitis C virus (HCV)
6. Women of childbearing potential will not be breastfeeding and will have a negative serum pregnancy test within 21 days of study drug administration as well as on Study Day -1
7. Women of childbearing potential (including peri-menopausal women who have had a menstrual period within 1 year of enrollment) must be using appropriate birth control (defined as a method with low failure rate, i.e., less than 1% per year, when used consistently and correctly such as implants, injectables, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner) during the entire duration of study participation. Use of contraceptive medications is allowed during the study. Women who have undergone a total hysterectomy or are postmenopausal are eligible.
8. In the opinion of the investigator, the subject is capable of understanding and complying with the protocol
9. Subject is a non-smoker, i.e., has refrained from any tobacco usage, including smokeless tobacco, nicotine patches, etc. for 6 months before study entry
10. Subject's normal alcohol consumption does not exceed 3 units per day if male or does not exceed 2 units per day if female. Both male and female subjects will be permitted to consume no more than 2 units of alcohol per day throughout the study. (One unit of alcohol is equivalent to 1 ounce of hard liquor, or 4 ounces of wine, or 12 ounces of beer.)
11. Willing to forego other forms of experimental treatment during the study

Exclusion Criteria:

1. Subject is unwilling or unable to comply with the protocol during the study period or to cooperate fully with the investigator or the site personnel
2. Subject has a significant organ abnormality or disease
3. Subject is considering or scheduled to have any surgical procedure during the duration of the study
4. Subject has an active malignancy or history of solid, metastatic, or hematologic malignancy with the exception of basal or squamous cell carcinoma of the skin that has been removed
5. Subject has donated or lost more than a unit of blood within 30 days before screening
6. Subject has a positive qualitative urine drug test at screening or an abnormal blood alcohol test (≥ 10mg/dL) on Study Day -1
7. Subject has received any other investigational drug or investigational biologically derived pharmaceutical agent within 60 days before screening
8. Subject has a history of seizure, chronic headache, viral encephalitis, or clinically significant infection (including viral) in the 14 days before dosing
9. Subject is receiving any concomitant medication requiring a prescription, except for contraceptives
10. Use of OTC preparations, herbal remedies or nutritional supplement (other than calcium and vitamin D) within the 7 days before study drug administration
11. Subject has ongoing drug abuse/dependence (including alcohol); or recent history (over the past 5 years) of, or treatment for, alcohol or drug abuse
12. Subject has a significant allergy to food or drugs
13. Currently symptomatic seasonal allergies, or history of anaphylaxis, asthma, dermatographism or eczema
14. Subject has any condition(s) that in the investigator's opinion would warrant exclusion from the study or prevent the subject from completing the study
15. Subject is unable to understand spoken and/or written English or any other language in which a certified translation of the informed consent is available

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events and serious adverse events through the end of the study. | 6 months

SECONDARY OUTCOMES:
The determination of pharmacokinetic (PK) parameters and immunogenicity of MGAWN1. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL Phase 1 Unit, Baltimore, Maryland, United States